CLINICAL TRIAL: NCT02991105
Title: Epidemiology of Cancer After Solid Organ Transplantation - EpCOT Study
Acronym: EpCOT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Adnan Sharif, Consultant Nephrologist, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: EpCOT
Record Dates: First submitted 2016-12-01; First posted 2016-12-13 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Malignancy
Keywords: Malignancy; Cancer; Organ Transplantation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Solid organ transplant recipients: National cohort = 85,410 solid organ transplant recipients receiving their transplant between January 1st 1985 to December 31st 2015

SUMMARY:
Cancer remains a major cause of morbidity and mortality post solid organ transplantation. While mortality from the other leading causes of death post-transplantation (e.g. cardiovascular disease and infection) is declining, mortality from cancer post-transplantation is increasing. This is due to both general and transplant-specific risk factors that combine to increase risk for cancer compared to the general population. However, there is a shortage of research exploring cancer epidemiology post solid organ transplantation in the UK. This is essential to guide clinicians and for counselling patients regarding expectations and outcomes after developing cancer post-transplantation. This is especially important as the aetiology, pathophysiology and outcomes of cancer post-transplantation may differ from the general population.

Available data registries in the UK separately contain valuable cancer and transplant-specific data that can be combined to explore cancer epidemiology post-transplantation more comprehensively, which can be directly translated into patient benefit by utilizing transplant-specific data (rather than translating from general population or non-UK patient demographics).

The purpose of this project is to combine existing data resources to link up the complete patient journey for solid organ transplant recipients nationally and focus on the entire spectrum of cancer from incidence to mortality.

DETAILED DESCRIPTION:
Solid organ transplantation is associated with an increased incidence of cancer versus the general population, and broadly on par with comparable immune deficiency states such as HIV/AIDS. The aetiology of cancer post-transplantation is primarily due to the burden of immunosuppression that is compulsory for all transplant patients to prevent allograft rejection. Skewed standardised incidence ratios are observed for cancer post-transplantation compared to the general population, with preponderance for cancers with a strong viral component. The literature on cancer-related mortality after transplantation is scarce, but again disparate mortality risk has been documented comparing solid organ transplant recipients to the general population.

There is a shortage of UK-specific data to guide transplant clinicians on how best to deal with cancer. This is important as countries differ with regards to ethnic demographics and post-transplant immunosuppression protocols, both of which are important confounders to translate data from other transplant cohorts. Collett and colleagues have previously published registry data of cancer incidence in British transplant recipients (by linking UK Transplant Registry to various national cancer registries) for a cohort transplanted between 1980 and 2007. They found similarities but also important differences between cancer incidence in a British solid organ recipient cohort versus registry data from Sweden, Finland, Canada and the United States. Importantly, the relevance of this data to the contemporary solid organ transplant cohort is unclear, as immunosuppression protocols have evolved since 2007 to a predominantly tacrolimus-based regimen since publication of the SYMPHONY study in 2007. No subsequent analysis has been done to determine the impact of tacrolimus introduction into cancer occurrence post-transplantation in the UK.

Previous work has analysed cancer-related mortality in the UK, providing data on site of cancer-related mortality and stratifying analysis along demographic factors such as age, gender and/or ethnicity that are relevant to the British population. This analysis linked two different national data resources from the study by Collett and colleagues - Hospital Episode Statistics and the Office for National Statistics. It demonstrated the crude cancer-related mortality rate in England (between 2001 and 2012) was 361 cancer-related deaths per 100,000 person years (compared to 424 and 416 for cardiovascular- and infection-related deaths respectively). Of note, cancer-related mortality within the first year post kidney transplantation (7.4%) has been shown to rise in incidence with increasing time post-transplantation (22.0% beyond the first year post kidney transplantation and second leading cause of death).

This previous work has identified the strengths and limitations of utilising such data resources. One of the major limitations with registry data is the absence of important and relevant information that can confound the data, which can be overcome by linking data between registries. For example, previous analyses identified kidney cancer accounted for over half of all cancer-related mortality for kidney transplant recipients with a history of pre-transplant cancer. However, the limitation of that data was the inability to probe this association further for a number of important issues; 1) location of kidney cancer (whether native or transplant kidney), 2) whether pre-transplant cancer was kidney-related, and 3) time on dialysis pre-transplant (which is a strong risk factor for acquired cystic renal disease and malignant transformation). While this information was unavailable in isolated data sets, such information is contained within other national data resources and could be combined by data linkage to create a broad and comprehensive epidemiological resource.

Data or record linkage has been defined as "a process of pairing records from two files and trying to select the pairs that belong to the same entity." Cancer data is not routinely collated by transplant centers and there is no robust mechanism to explore cancer epidemiology data post solid organ transplantation through the UK Transplant Registry. However, linking information to other existing data registry resources will facilitate such analysis. This is an under-researched area within both transplant and cancer communities, but increasingly important due to the increasing incidence and prevalence of cancer post solid organ transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Solid organ transplant recipient, transplant performed in England

Exclusion Criteria:

* Transplant performed in Scotland, Wales or Northern Ireland
* Any living transplant recipient who wishes to opt-out of the anonymised record linkage (contact study lead: central contact person)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 85,410 solid organ transplant have been performed in England between 01/01/1985 and 31/12/2015.
Sampling Method: Non-Probability Sample
Enrollment: 85410 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Cancer-related mortality after solid organ transplantation | 1985-2016 cohort
  To compare observed and expected risks of specific causes of deaths, in particular cancer-related death, by linking the UKTR with the national death registry to obtain underlying causes of death and determine factors related to increased risk of specific causes of death post-transplantation. General population mortality rates will be used to calculate expected number of deaths from specific causes and identify subgroups of post-transplant patients (e.g. age, sex, transplant centre, organ type, etc.) at excess risk compared with expected risk.
  Investigate survival and causes of death after cancer in post-transplant patients versus individuals from the general population with a similar de novo cancer of the same age, sex, and calendar year of diagnosis.

SECONDARY OUTCOMES:
Risk for cancer after solid organ transplantation | 1985-2016 cohort
  Compare observed and expected risks of specific cancer types post-transplantation by linking the UKTR with the national cancer registry to obtain observed numbers of cancers and determine factors related to increased risk of specific types of cancer. General population cancer incidence rates will be used to calculate expected numbers of cancers of specific type and identify subgroups of post-transplant patients at excess risk of specific cancers compared with expected.
Associated morbidity after developing cancer after solid organ transplantation | 1985-2016 cohort
  Estimate risk of morbidity requiring hospitalisation both generally and that associated with development of post-transplantation cancer by linking the UKTR with Hospital Episode Statistics (HES). Risk of hospital admissions and procedures (e.g. surgery) for specific morbidities will be investigated. We will calculate expected risks for specific conditions requiring hospitalisation, enabling identification of specific subgroups of post-transplant patients at excess risk compared with expected.
Risk prediction for cancer after solid organ transplantation | 1985-2016 cohort
  Machine learning utilising patient level data from linked registries to risk stratify solid organ transplant recipients at risk for cancer

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - University of Birmingham, Birmingham

IPD SHARING:
Plan to Share IPD: No